CLINICAL TRIAL: NCT02682199
Title: Prospective Evaluation of Patient-Reported Xerostomia After Whole Brain Radiation
Brief Title: Prospective Evaluation of Patient Reported Xerostomia After Whole Brain Radiation
Acronym: NRR
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1540
Record Dates: First submitted 2016-01-20; First posted 2016-02-15 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Whole Brain Radiation: Patients scheduled to receive whole brain radiation with or without chemotherapy/targeted therapy.

SUMMARY:
The goal of this prospective observational study is to investigate whether whole brain radiation leads to measurable xerostomia from parotid gland toxicity.

DETAILED DESCRIPTION:
The parotids have not been traditionally considered an organ at risk / avoidance structure in whole brain radiation. However, patients receiving whole brain radiation sometimes complain of dry mouth. Investigators hypothesize that standard whole brain radiation fields cause an acute measurable increase in xerostomia at one month post-radiation, and that the severity of xerostomia is related to the dose received by the parotids. In this study, investigators will use the validated University of Michigan Xerostomia Questionnaire to prospectively collect baseline and post-radiation xerostomia scores up to 6 months after treatment. The radiation dose to the parotids will be evaluated to assess whether there is a dose-toxicity relationship. Investigators anticipate a total accrual of 60 patients with a goal of 48 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients to be treated with whole brain radiation in 10-15 fractions to a total dose of 25-37.5 Gy for a diagnosis of brain metastases from any disease site or as prophylaxis in the treatment of potentially subclinical intracranial disease (e.g. from small cell lung cancer).
* Has not had prior radiation that would have exposed the parotids to a significant (estimated >10 Gy mean parotid dose) level of radiation within the past one year. Patients receiving prior stereotactic radiosurgery for brain metastasis are eligible for inclusion in this trial as this form of radiation is highly conformal and exposes the parotids to minimal (estimated <1 Gy) radiation.
* Greater than or equal to 18 years of age (no upper age limit).
* Informed consent obtained.

Exclusion Criteria:

* Patients receiving whole brain radiation without the use of a CT-based planning simulation.
* Patients who are on medications known to cause dry mouth, such as anticholinergics.
* Physically unable to communicate by paper or phone to complete the study survey.
* Prisoners.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing whole brain radiation treatment at Lineberger Comprehensive cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Measureable acute increase in xerostomia | baseline to 1 month post-treatment

SECONDARY OUTCOMES:
Association of degree of change in xerostomia score and the radiation dose received by the parotid glands | baseline to 1 month post-RT
Effect of whole brain radiation on the time course of xerostomia | baseline and four post-radiation time points (procedure, 1 month post-RT, 3 months post-RT, 6 months post-RT).

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Wang, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org/